CLINICAL TRIAL: NCT04557007
Title: Drug Concentration Monitoring of Pembrolizumab in Treatment-naive Non-Small Cell Lung Cancer Patients
Brief Title: Drug Concentration Monitoring of Pembrolizumab in Non-Small Cell Lung Cancer Patients
Acronym: Oncomabs
Status: Terminated | Type: Observational
Why Stopped: Difficulty recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Ragnhild Nome, Principal Investigator, Oslo University Hospital
Other Study IDs: 2017/9660
Record Dates: First submitted 2020-09-02; First posted 2020-09-21 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and full blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment-naive NSCLC patients: Treatment-naive NSCLC patients receiving immunotherapy (pembrolizumab) alone or in combination With chemotherapy divided in groups based on treatment administered. Clinical information will be gathered at start of treatment and at evaluations every 3rd month.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Drug trough-level will be measured in patients on Pembrolizumab with or without additional chemotherapy in routine care.

SUMMARY:
This observational study explores associations between drug trough-levels and clinical outcomes in Non Small Cell Lung Cancer (NSCLC) patients treated with immunotherapy (pembrolizumab) either alone or combined with chemotherapy. Through-levels of pembrolizumab will be examined in blood samples collected during the first-line treatment period. In addition T-cell responses in peripheral blood and anti-drug antibodies will be monitored. Results of drug trough-levels and T-cell responses will be linked to clinical outcome. 250 patients with NSCLC will be enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be > 18 years and must voluntary sign an informed consent
* Treatment-naïve patients with advanced NSCLC receiving immunotherapy alone (pembrolizumab) or combined with chemotherapy

Exclusion Criteria:

* Any anti-cancer therapy < 6 months prior to study start
* Radio- or chemotherapy against lung cancer <2 years before study start
* Previous treatment with immunotherapy
* Patients with mutations with specific treatment (i.e. EGFR, ALK, Ros1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients With Advanced disease elligible for routine treatment With immunotherapy alone or in combination With chemotherapy.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Objective response | 3 months
  Radiological response (Partial response/stable disease/Complete response)

SECONDARY OUTCOMES:
Adverse events | 2 years
  Adverse events >= 3
PD-1 Expression on CD-8 T-cells | First 3 months
  Proliferation of PD-1 Expression CD-8 T-cells
Overall survival | 5 years observation
  Overall survival related to drug trough-level
Progression-Free survival | 1 year
  Radiological evaluation

OTHER OUTCOMES:
Pembrolizumab clearance | 3 months
  mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Ragnhild Nome, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- St Olavs University Hospital, Trondheim, Norway